CLINICAL TRIAL: NCT03150784
Title: Brain Plasticity and Motor Skill Competence Development in Young People With Development Coordination Disorder
Brief Title: Rhythmic Motor Learning in Children With Developmental Coordination Disorders
Acronym: EPIC2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: University of Oxford (Other); National University of Ireland, Maynooth (Other)
Responsible Party: Principal Investigator, Helen Dawes, Professor, Movement Science Group, Faculty of Health and Life Sciences, Oxford Brookes University, Oxford Brookes University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 161033
Record Dates: First submitted 2017-04-04; First posted 2017-05-12 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Developmental Coordination Disorder
Keywords: Motor Learning; Coordination; Children; Motor Skills Disorders; Movement
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: Measures taken at Baseline (0 weeks), Post Intervention (6-7 weeks), and follow up (12 weeks)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motor coordination difficulties (Experimental): Type: Experimental main
  EPIC club: 60min session / 2 times weekly / 7 weeks
  Interventions: Other: EPIC Club
- Non motor coordination difficulties (Other): Type: Experimental comparator
  EPIC club: 60min session / 2 times weekly / 7 weeks
  Interventions: Other: EPIC Club

INTERVENTIONS:
Other: EPIC Club — Weekly exercise gym sessions. Participants will start with a warm-up of 20-25 mins cardiovascular training either doing cycling, treadmill running or cross-training. The remainder of the session consists of strength/resistance and weight-training involving leg press, leg extensor, pull downs, kettle bells, dumbbells. In addition to the above, a novel rhythmical stepping task will be performed over 10 mins.

SUMMARY:
The importance of play and physical activity include many benefits on positively improving health and well-being, enhancing children's and young people's thinking and performance in school, improving their sleep and enabling confidence and skill building. However, some children find it hard to learn and perform motor skills, and are at risk of decreased participation in sports and physical activity and subsequently decreased physical fitness and overall health and well-being.

Previous studies from the research group have explored the impact and recovery following acute exercise at different intensities in children and adolescents with and without movement difficulties. Following this, a pathway promoting physical activity and engagement has been successfully established within schools for those with and without movement difficulties. Taking the previous studies further, we want to specifically focus on the children's performance and learning of a sporting skill, such as stepping, and the associated brain activity changes, using available high resolution imaging techniques. This will help us understand how these children perform and learn motor and sporting skills. Evidence obtained from imaging alongside measures of movement has helped the development of optimal therapeutic approaches for other conditions such as stroke and Parkinson's and will help us to develop approaches to help children best learn motor skills and hence gain confidence in performing sporting activities.

DETAILED DESCRIPTION:
Children with poor motor skill acquisition and execution despite having opportunity for learning, are now described as having developmental coordination disorder (DCD). There is a prevalence of 5-6% of young people who have normal intelligence who meet this category who have problems affecting their activities of daily living (ADL's). Young people with lower motor skills are one of a number of conditions affecting children identified by the Chief Medical Officer as requiring an improved evidence base for management. Poor motor skill acquisition and execution, whereby skills remain substantially lower than expected despite opportunities for learning; interferes with participation in academic, sporting and leisure activities. Motor performance is slower and of poor quality; and children may have difficulties learning all kinds of motor skills including sporting activities. Importantly people with poor motor skill acquisition and execution can fail to establish the fundamental movement skills and literacy required to integrate in physical pursuits, such as sport, and become exposed to long-term conditions associated with inactivity. Motor sporting skills can be learnt if trained, but difficulties in performing and learning skills persist into adulthood.

Brain imaging during rhythmic motor tasks which are essential in day-to-day (non-)sporting activities, have established that children with poor motor skill acquisition and execution show differences to healthy controls in grey and white matter functional connectivity and in cortical activation patterns during performance of simple movement tasks . Provisional evidence suggests that individuals with poor motor skill acquisition and execution utilise activation processes when learning motor tasks that are more controlled and require extra processing demands, but a systematic review of neural correlates of those with poor motor skill acquisition and execution concludes that data is scarce and more studies are needed. Performance of motor tasks requires a balance between automatic and controlled processes that is dependent upon the demands of the task and the capabilities of the individual. Young people need to be able to consider their environment when performing a sport rather than just thinking about the skill, so that they can work out where the best place to kick a ball on a football pitch is, not just kick the ball. Typically developing (TDC) children acquire motor skills either implicitly or explicitly by observing and imitating other children and adults or by trial and error. Acquisition of motor tasks requires plasticity in the nervous system with improvements in motor performance underpinned by a move from cortically controlled mechanism, towards more automatic performance, freeing up cortical resources. The ability to automate certain parts of motor skills allows the execution of tasks in more complex environments. Provisional evidence suggests that people with poor motor skill acquisition and execution may learn motor skills in a more controlled manner and have a reduced ability to move automatically. To date no studies have explored the brain changes underpinning fundamental motor skills attainment over a training period in people with poor motor skill acquisition and execution.

The main aim contribute evidence towards describing motor performance in relation to brain structure and functioning in children with lower motor skills and DCD,. This study proposes to test both the feasibility and determine the extent of the impact of learning a novel coordination task on motor performance and brain structure and functioning in children with DCD to inform a full-scale trial of skill acquisition.

ELIGIBILITY:
Inclusion Criteria:

* 12-15 years old children (year 9 students only) with normal intelligence in the lowest quartile of fitness (30 with poor motor skill acquisition and performance affecting daily functioning, 30 who score in the lower 25% of fitness measures without poor motor skill acquisition and execution).

Exclusion Criteria:

* Behavioural/intellectual issues that prevent safe participation or may put the participant, investigators and others at risk.
* Any contraindications to perform maximal exercise or physical training, as determined by the Physical Activity Health Questionnaire PARQ sent out to parents before screening.
* Children suffering from muscular/neurological degenerative conditions or with uncontrolled epilepsy/seizures (must be stable epilepsy/on medication for greater than 12 weeks).
* Surgical procedures in the previous 6 months.
* If there are any concerns regarding a child being able to participate safely, we will ask parents/guardians to contact the GP/paediatrician/physiotherapist.
* MRI Scanner: children with metal objects due to surgery or dental care cannot partake in the scanning part of the research.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Novel Stepping Task (assessing change over time) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Rhythmic stepping task measuring coordination
Functional Near-Infra red Spectroscopy (FNIRs) (assessing change over time) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Monitoring haemodynamic change of the cortex

SECONDARY OUTCOMES:
Physical Activity Audit (PAQ-A) (assessing change over time) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Questionnaire
Functional Magnetic Resonance Imaging (FMRI) (assessing change over time) | Baseline - change from baseline 6-7 weeks
  Monitoring change in brain activity
Movement Assessment Battery for Children 2 | Baseline
  Measuring Motor Coordination
Inertial Measurement Unit (IMU) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Accelerometry Gait Analysis
Child Health Utility Questionnaire 9D (assessing change over time) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Questionnaire
Harter's Self-Perception Profile for children (assessing change over time) | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  Questionnaire
Axivity AX3 Accelerometer | Baseline - change from baseline 6-7 weeks - change from baseline 12 weeks
  7 Day physical activity measurement

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Cherwell School, Oxford, OXON
  - Clinical Exercise Rehabilitation Unit, Oxford, OXON
  - Oxford Brookes University, Oxford, OXON
  - Cheney School, Oxford, OXON
  - Wheatley Park School, Oxford, OXON

IPD SHARING:
Plan to Share IPD: No
As per ethical outline, data will not be stored in a shared repository. All data will be stored in an anonymised format on site. Data access requests should be made to the principle investigator in writing which will be discussed in the data monitoring committee meetings.

REFERENCES:
- [Derived] Liu YC, Esser P, Weedon BD, Springett D, Joshi S, Tsou MH, Wang RY, Dawes H. Knee joint position sense and kinematic control in relation to motor competency in 13 to 14-year-old adolescents. Ital J Pediatr. 2024 Sep 29;50(1):200. doi: 10.1186/s13052-024-01765-z. PMID 39343969
- [Derived] Inacio M, Esser P, Weedon BD, Joshi S, Meaney A, Delextrat A, Springett D, Kemp S, Ward T, Izadi H, Johansen-Berg H, Dawes H. Learning a novel rhythmic stepping task in children with probable developmental coordination disorder. Clin Biomech (Bristol). 2023 Feb;102:105904. doi: 10.1016/j.clinbiomech.2023.105904. Epub 2023 Feb 3. PMID 36764101